CLINICAL TRIAL: NCT00006256
Title: Concurrent Taxol (Paclitaxel) and Definitive Breast Radiation Therapy in Early Stage Breast Cancer Following Four Cycles of Adriamycin/Cytoxan Chemotherapy
Brief Title: Paclitaxel Plus Radiation Therapy in Treating Women With Stage II or Stage III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU2199
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: paclitaxel — Patients receive paclitaxel IV over 3 hours every 21 days for 4 courses beginning 3 weeks after completion of the last doxorubicin and cyclophosphamide adjuvant regimen.
Procedure: adjuvant therapy — doxorubicin and cyclophosphamide adjuvant regimen
Radiation: radiation therapy — Patients also undergo concurrent radiotherapy 5 days a week for approximately 6-7 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining paclitaxel with radiation therapy may kill more tumor cells.

PURPOSE: This trial is to study the effectiveness of concurrent administration of chemotherapy and radiation therapy in treating women who have stage II or stage III breast cancer by examining the complications and cosmetic effects.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of concurrent paclitaxel and breast radiotherapy in women with stage II or III breast cancer who have had primary breast conserving surgery and adjuvant chemotherapy.
* Assess the cosmetic results of breast conservation after this treatment in these patients.
* Determine the pulmonary toxicity of this regimen in these patients.

OUTLINE: Patients receive paclitaxel IV over 3 hours every 21 days for 4 courses beginning 3 weeks after completion of the last doxorubicin and cyclophosphamide adjuvant regimen. Patients also undergo concurrent radiotherapy 5 days a week for approximately 6-7 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 month, every 3 months for 1 year, every 6 months for the next 5 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study over 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Stage II or III invasive breast cancer
* Prior breast conserving surgery (lumpectomy or quadrantectomy) with ipsilateral axillary lymph node dissection required
* No prior contralateral breast cancer
* No metastatic disease
* Prior ductal carcinoma in situ or lobular carcinoma in situ of the breast allowed unless treated with radiation or chemotherapy
* Doxorubicin and cyclophosphamide adjuvant chemotherapy completed within past 3 weeks
* Candidate for definitive radiotherapy
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm3
* Granulocyte count at least 2,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT/AST no greater than 1.5 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No concurrent poorly controlled ischemic heart disease or congestive heart failure
* LVEF at least 45% by MUGA scan or echocardiogram

Pulmonary:

* No concurrent severe chronic obstructive or restrictive pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No concurrent severe medical or psychiatric illness
* No concurrent severe diabetes mellitus
* No other prior malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix treated with local excision

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent filgrastim (G-CSF)

Chemotherapy:

* See Disease Characteristics
* Prior tamoxifen allowed
* No concurrent tamoxifen

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiation to the breast

Surgery:

* Recovered form prior surgery

Other:

* No concurrent adjuvant therapy on another clinical trial

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2000-06-08 (Actual); Primary Completion 2005-11-30 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of concurrent paclitaxel and breast radiotherapy | Followed every 3 months for 1 year
  Ability to deliver appropriate doses of radiation therapy within the appropriate time course
chemotherapy dose achieved during concurrent Taxol and radiation therapy. | Followed every 3 months for 1 year

SECONDARY OUTCOMES:
Cosmetic outcome based upon established descriptive parameters: excellent, good, fair, and poor. | 1 year
  These parameters will be assessed by medical and radiation oncology. We expect at least a > 60% completion rate with this treatment, which translates into confidence limits of 46% to 74% when 40 patients are investigated.
Pulmonary function | 1 year
  Combined treatment impact on pulmonary function. Evidence of pulmonary toxicity demonstrated by a reduction in DLCO (Diffusing Capacity of the Lung for Carbon Monoxide).
Survival | 5 years
  Patients followed for long term survival for at least 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Lyons, MD, Study Chair — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (9):
- United States (9):
  - UH-CantonMercy, Canton, Ohio
  - UH-Geauga, Chardon, Ohio
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - UH-Monarch, Mayfield Heights, Ohio
  - UH-LUICC, Mentor, Ohio
  - UH-Southwest, Middleburg Heights, Ohio
  - UH-Chagrin Highlands, Orange, Ohio
  - UH-Green Road, South Euclid, Ohio
  - UH-Westlake, Westlake, Ohio